CLINICAL TRIAL: NCT02255240
Title: LEVEL UP: Leveraging Electronic Videogames for Exercise and Leisure: Understanding Preferences of Breast Cancer Survivors
Brief Title: LEVEL UP: Video Games for Activity in Breast Cancer Survivors
Acronym: LEVEL UP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Relinquished grant funding due to receipt of another incompatible grant
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-0240; 1K07CA175141-01A1 (NIH)
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer; Obesity
Keywords: breast cancer; cancer; survivorship; cancer survivor; physical activity; video game; women; women's health
MeSH Terms: conditions — Breast Neoplasms; Obesity; Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical activity intervention (Experimental): This arm will receive the physical activity intervention, which consists of three individual meetings, weekly brief counseling phone calls for 6 weeks, and provision of a video game console with three active video games.
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — Participants will receive counseling on self-regulatory skill building that has been adapted to complement the video games used. We anticipate that the games used will consist of fitness, sports, and dance games and will be played on a Wii U console. The games played will be chosen by each participant from a pool of potential appropriate games.

SUMMARY:
The purpose of this study is to test an intervention that uses home console video games to encourage increased physical activity among postmenopausal breast cancer survivors.

DETAILED DESCRIPTION:
This research project includes qualitative and quantitative formative research leading to a randomized controlled feasibility trial of a video game-based physical activity intervention. First, we will investigate exercise protocols implemented over 6 weeks in 20 breast cancer survivors. We will choose a console and six games for inclusion in the trial, based on measured energy expenditure and enjoyment. We will create refined exercise protocols using these games and insights from participants. Second, we will test an intervention that uses active video games for implementation of motivating exercise and provision of behavioral tools (e.g., tracking of progress towards goals). Participants in a pre-pilot trial (N = 10) will receive weekly brief telephone counseling over 6 weeks. Feasibility measurement will include attrition, self-reported acceptability, and objective measures of video game play taken from game console data.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 45 - 75
* Diagnosed with breast cancer within the past 10 years

Exclusion Criteria:

* Chemotherapy or radiation treatment in the past six months
* Surgery in the past six months
* Evidence of disease recurrence
* Unable to read and understand English
* Unable to see a TV screen from several feet away
* Unable to find transportation to the study location
* No Internet access in the home (only for intervention portion of the study)
* Participant is active (60 minutes of moderate-vigorous intensity activity per week or more)
* BMI is under 18.5 kg/m2 or over 40 kg/m2
* Participant reports psychological issues that would interfere with study completion. Examples will be provided to illustrate potential psychological issues, such as dementia or schizophrenia.
* Inadequate performance on Senior Fitness Test, indicating inability to engage in video game exercise procedures (total score < 9 out of 12)
* Report a heart condition, chest pain during periods of activity or rest, loss of consciousness, etc. on the Physical Activity Readiness Questionnaire (PAR-Q), unless cleared by their physician
* Unable to walk, jump, and jog as may be required by some games (self-report)
* Report current symptoms of alcohol or substance dependence
* Plans to move away from the Galveston-Houston area or to be out of town for more than 1 week during the study period
* Unwillingness to report drugs taken for comorbidities such as hypertension or diabetes
* Stroke, hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
* Report a history of orthopedic complications that would prevent optimal participation in the physical activities prescribed (e.g., heel spurs, severe arthritis)
* Clinical judgment concerning safety
* Currently participating in a physical activity or weight program/research study
* Currently pregnant or nursing
* No TV is available in the participant's home
* Currently on a weight loss diet or has lost more than 5% body weight in the previous 6 months
* Current smoker
* Game console to be used in the study is already available in the home
* Another member of the household is a participant or staff member on this trial

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity from baseline to 6 weeks | 6 weeks
  Minutes of moderate-vigorous physical activity measured over a 7 day period

SECONDARY OUTCOMES:
Change in physical fitness from baseline to 6 weeks | 6 weeks
  We will use a six minute walk test to measure fitness
Change in weight from baseline to 6 weeks | 6 weeks
  Weight will be measured using a calibrated scale
Change in motivation from baseline to 6 weeks | 6 weeks
  We will measure autonomous motivation (intrinsic, integrated, identified, etc.) specific to physical activity
Change in body function from baseline to 6 weeks | 6 weeks
  We will use the Senior Fitness Test to measure strength and body function
Change in quality of life from baseline to 6 weeks | 6 weeks
  We will use the Functional Assessment of Cancer Therapy - Breast measure to quantify quality of life

OTHER OUTCOMES:
Number of participants who drop out of the study from baseline to 6 weeks | 6 weeks
  We will investigate the number of participants who drop out of the intervention group in comparison to similar studies
Acceptability | 6 weeks
  We will measure acceptability of the intervention components and tools using validated self-report measures and qualitative interviews/focus groups
Number of participants who report adverse events | 6 weeks
  We will inquire about potential adverse events during counseling calls and assessment visits. Discrete events will be summed, and the number of participants with events will be summed.
Adherence | 6 weeks
  We will use objective measures to investigate adherence to game play protocols (console logs, automatic postings to the console social network, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Lyons, PhD, MPH, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States